CLINICAL TRIAL: NCT06111547
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, Single and Multiple Oral Doses Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of TAK-279 in Healthy Chinese Subjects
Brief Title: A Study of TAK-279 in Healthy Chinese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TAK-279-1005
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: TAK-279 30 mg (Experimental): Participants will receive a single dose of TAK-279 30 milligram (mg) oral tablet on Day 1 followed by Day 6 to Day 19 once daily under fasted condition.
  Interventions: Drug: TAK-279
- Cohort 2: TAK-279 60 mg (Experimental): Participants will receive a dose of TAK-279 60 mg (2*30mg) oral tablets on Day 1 followed by Day 6 to Day 19 once daily under fasted condition.
  Interventions: Drug: TAK-279
- Cohort 1 and 2: Placebo 30 mg or 60 mg (Placebo Comparator): Participants will receive TAK-279 30 mg or 60 mg (2*30mg) matching placebo oral tablets on Day 1 followed by Day 6 to Day 19 once daily under fasted condition.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-279 — TAK-279 oral tablet.
  Arms: Cohort 1: TAK-279 30 mg; Cohort 2: TAK-279 60 mg
Drug: Placebo — TAK-279 30 mg or 60 mg (2*30mg) matching placebo tablet.
  Arms: Cohort 1 and 2: Placebo 30 mg or 60 mg

SUMMARY:
The main aim of this study is to find out how the body of a healthy Chinese adult processes TAK-279 (pharmacokinetics). Other aims are to learn about side effects and how well TAK-279 is tolerated when given to healthy Chinese Adults. Participants will receive either TAK-279 or a placebo on Day 1 and from Day 6 to Day 19. Blood samples will be taken at different timepoints throughout the study participation. Participants will need to adhere to certain lifestyle restrictions during the study. This also includes eating and drinking restrictions.

During the study, participants will need to stay at the clinic for 25 days.

ELIGIBILITY:
Inclusion criteria:

* Participant is willing to participate and is capable of giving informed consent.
* Healthy, male or female participants of Chinese descent 18 to 45 years of age, inclusive, at the time of informed consent.
* Female participants meets the following contraception requirements: A surgically sterile female participant; or a female participant of nonchildbearing potential with laboratory confirmation of postmenopausal status (that is follicle-stimulating hormone levels greater than [>] 40 milli-international units per milliliter [mIU/mL]); or, if sexually active with a non-sterilized male partner, a female participant who agrees to use a highly effective method of contraception from the signing of informed consent throughout the duration of the study and for 10 days after the last dose. Male participants must agree to comply with effective contraceptive requirements.
* Body mass index greater than or equal to (>=) 18.0 kilogram per meter square (kg/m^2) and less than or equal to (<=) 28.0 kg/m^2 at the screening visit.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms [ECGs], as deemed by the principal investigator (PI) or designee, including the following:

  * Seated blood pressure (BP) (systolic BP/diastolic BP) >=90/50 millimeters of mercury (mmHg) and <=140/90 mmHg at the screening visit.
  * Seated heart rate or pulse is >=50 beats per minute (bpm) and <=100 bpm at the screening visit.
  * ECG findings are considered normal or not clinically significant by the PI or designee at the screening visit.
* Participant must be willing and able to understand and fully comply with all study procedures and must be available for the duration of the study.

Exclusion criteria:

* Site personnel or their family.
* History or presence of clinically significant medical or psychiatric condition or disease.
* History of any illness or condition that might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* History of allergy to study drug or any of its components.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
* Clinical laboratory values at the time of screening or at check-in:

  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) >1.5 * the upper limit normal (ULN).
  * Creatine phosphokinase (CPK) > the ULN.
  * Hemoglobin <11.0 grams per deciliter (g/dL) (<110.0 gram per liter [g/L]).
  * Absolute neutrophil count <1.8*10^9/liters (L) (<1800 per cubic millimeter [/mm^3]).
  * Absolute lymphocyte count <0.8*10^9/L (<800/mm^3).
  * Platelet count <100*10^9/L (<100,000/mm^3).
* A participant with out-of-range values may have the test repeated once at each time point (screening or check-in) and the participant may be enrolled if the repeated values are within protocol-specified ranges.
* Ingestion of Seville orange- or grapefruit-containing foods or beverages within 7 days prior to check-in.
* History of alcohol abuse or drug/chemical abuse within 2 years prior to check-in.
* Continuous smoker who has used nicotine- or tobacco-containing products within 1 month prior to the first dosing based on participant self-reporting.
* Female participants who have a positive pregnancy test result at the screening visit or at check-in, are planning to become pregnant during the study or are lactating.
* Positive results for urine drug test at the screening visit or at check-in.
* Herpes infections:

  * Participants has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at screening or check-in.
  * Participants has a history of serious herpetic infection that includes any episode of disseminated disease, multi-dermatomal herpes zoster virus, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
* Positive results for non-herpetic viral diseases at the screening visit:

  * Participant has presence of hepatitis C virus (HCV) antibody or a positive confirmatory test result for HCV RNA (Ribonucleic acid) test or polymerase chain reaction (PCR).
  * Participant has presence of positive result for hepatitis B surface antigen, presence of hepatitis B virus deoxyribonucleic acid, or positive anti-hepatitis B core antibody without concurrent positive hepatitis B surface antibody.
* Participant has positive results for human immunodeficiency virus.
* Positive results for Tuberculosis (TB) at the screening visit:

  * The participant has a history of active TB infection, regardless of treatment status.
  * The participant has signs or symptoms of active TB (including but not limited to chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the investigator.
  * The participant has evidence of latent TB as evidenced by a positive QuantiFERON-TB Gold (QFT) result or tuberculosis-specific enzyme-linked immunospot assay (T-Spot) OR 2 indeterminant QFT results or 2 borderline T-Spot results.
  * The participant has had any imaging study during or 6 months prior to screening, including x-ray, chest computed tomography, magnetic resonance imaging, or other chest imaging suggesting evidence of current active or a history of TB.
* Positive result for Coronavirus disease 2019 (COVID-19) PCR test at the screening visit.
* Prior and concomitant therapy:

  * Participants who received a live or live-attenuated vaccine in the 60 days prior to study drug administration. Administration of nonlive-attenuated vaccines or boosters for COVID-19 (for example [eg,] RNA-based vaccines, inactivated adenovirus-based vaccines, protein-based vaccines) in the 14 days prior to first dosing. The study site should follow local guidelines related to COVID-19.
  * Use or intent to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including CYP3A4 and/or P-glycoprotein (P-gp) inhibitors or inducers and St. John's wort, within 30 days prior to check-in.
  * Use or intent to use any prescription medications/products or over-the-counter (OTC) medications within 14 days prior to check-in.
  * Use or intent to use any nonprescription medications/products including phyto-therapeutic/herbal/plant-derived preparations within 14 days prior to check-in
* Donation of blood or significant blood loss within 56 days prior to study drug administration. Plasma donation within 7 days prior to the first dosing.
* Participation in another clinical study and having received its study drug within 30 days or 5 elimination half-lives prior to study drug administration. The 30-day or 5 elimination half-lives window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-08-04 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Time Curve From Time 0 to the Time t (AUC0-t) of TAK-279 | Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  AUC0-t of TAK-279 in plasma will be assessed.
Area Under the Concentration-time Curve From Time 0 To Infinity (AUC0-inf) of TAK-279 | Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  AUC0-inf of TAK-279 in plasma will be assessed.
Maximum Observed Plasma Concentration (Cmax) of TAK-279 | Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Cmax of TAK-279 in plasma will be assessed.
Area Under the Concentration-Time Curve During a Dosing Interval (AUCtau) of TAK-279 | Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  AUCtau of TAK-279 in plasma will be assessed.
Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of TAK-279 | Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Cmax,ss of TAK-279 in plasma will be assessed.

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events of Special Interest (AESI) | From start of study drug administration up to follow-up (up to Day 36)
  Number of participants with TEAEs, serious TEAEs and AESI will be reported.
Number of Participants With Clinically Significant Changes in 12-Lead Electrocardiogram (ECG), Vital Signs and Clinical Laboratory Parameters | From start of study drug administration up to follow-up (up to Day 36)
  Number of participants with clinically significant changes in ECG, vital signs, and clinical laboratory parameters will be assessed. Clinical significance of ECG, vital signs, and clinical laboratory parameters will be determined at the investigator's discretion.
Area Under the Plasma Concentration-Time Curve From Time 0 To the Time 24 Hours (AUC0-24) of TAK-279 | Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
  AUC0-24 of TAK-279 in plasma will be assessed.
Terminal Elimination Rate Constant (Lambda z) of TAK-279 at Day 1 and Day 19 | Day 1 and Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Lambda z of TAK-279 in plasma will be assessed.
Terminal phase half-life (t1/2) of TAK-279 at Day 1 and Day 19 | Day 1 and Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  t1/2 of TAK-279 in plasma will be assessed.
Apparent Clearance (CL/F) of TAK-279 | Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  CL/F of TAK-279 in plasma will be assessed.
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of TAK-279 | Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Vz/F of TAK-279 in plasma will be assessed.
Time to Reach Peak Plasma Concentration (Tmax) of TAK-279 | Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Tmax of TAK-279 in plasma will be assessed.
Minimum Plasma Concentration (Cmin) of TAK-279 | Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Cmin of TAK-279 will be assessed.
Trough Concentration (Ctrough) of TAK-279 | Pre-dose on Day 17, Day 18 and Day 19
  Ctrough of TAK-279 will be assessed.
Time to Reach the Maximum Plasma Concentration at Steady State (Tmax,ss) of TAK-279 | Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Tmax,ss of TAK-279 will be assessed.
Total Body Drug Clearance at Steady State (CLss/F) of TAK-279 | Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  CLss/F of TAK-279 will be assessed.
Apparent Volume of Distribution at Steady State (Vss/F) of TAK-279 | Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Vss/F of TAK-279 will be assessed.
Average Plasma Concentration (Cavg) for TAK-279 | Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Cavg of TAK-279 will be assessed, calculated as AUC(tau)/tau. Tau is defined as length of dosing interval.
Percent peak-to-trough fluctuation (%FLUC) of TAK-279 | Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Percent peak-to-trough fluctuation will be assessed, calculated as 100%*([Cmax,ss-Ctrough]/Cavg) will be assessed.
Accumulation Ratio for Cmax (RA, Cmax) of TAK-279 | Day 1 and Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Accumulation ratio calculated from Cmax,ss at steady state and Cmax indicated a single dose will be assessed.
Accumulation Ratio for AUCtau (RA, AUCtau) of TAK-279 | Day 1 and Day 19: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose
  Accumulation ratio calculated from AUCtau at steady state and AUC0-24 indicated a single dose will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Huashan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/878f1c20e19f46a5?idFilter=%5B%22TAK-279-1005%22%5D